CLINICAL TRIAL: NCT00990483
Title: A Comparison of 15 and 30 Acquisition Angle Breast Tomosynthesis Mammography in the Visualization and Characterization of Breast Abnormalities
Brief Title: A Comparison of the 15 and 30 Acquisition Angle Breast Tomosynthesis Mammography for Breast Abnormalities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hologic, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 09-02
Record Dates: First submitted 2009-10-05; First posted 2009-10-06 (Estimated); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Tomosynthesis; 3D Mammogram; Diagnostic mammogram
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 3D investigational imaging (Experimental): patients returning with an area of interest will undergo investigational 3D imaging in 2 modes of imaging to the breast of interest and compare to the subjects standard of care imaging
  Interventions: Device: 3D mammograpgy system

INTERVENTIONS:
Device: 3D mammograpgy system — In addition to the standard care diagnostic imaging, all participants underwent two experimental acquisitions, in two projections (Cranio-Caudal and Mediolateral Oblique) on the breast of concern: one acquisition in Mode A (narrow angle acquisition) and one acquisition in Mode B (wide angle acquisition). The experimental imaging is compared to the standard of care imaging
  Other Names: Selenia Dimensions; Tomosynthesis

SUMMARY:
The purpose of this study is to conduct an initial investigation into whether an alternative method of using 3D imaging might offer accurate diagnostic performance at a reduced patient radiation exposure in comparison to conventional 2D screening and diagnostic mammography and conventional 2D + 3D imaging methods.

ELIGIBILITY:
Inclusion Criteria:

* Subject is female of any race and ethnicity
* Subject is at least 40 years old
* The screening and diagnostic mammograms were performed at the recruiting institution on a Hologic Selenia System
* Subject is categorized as BI-RADS 0 because if mass, density, or calcifications detected on the basis of screening or diagnostic mammography
* Subject will undergo study imaging within 30 days of standard of care imaging

Exclusion Criteria:

* Patients who are pregnant or think they may be pregnant
* Patients who are breast feeding
* Subjects unable or unwilling to undergo informed consent
* Subjects with breast implants

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2009-10; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
If the new imaging modes are successful, they will represent a method of reducing patient exposure for future imaging because they are designed to be used in 3D imaging only. | Fall 2010

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Farjardo, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States